CLINICAL TRIAL: NCT04920292
Title: A Phase 1, Bioavailability Study to Investigate the Pharmacokinetics, Safety and Tolerability of an Oxfendazole Tablet Formulation in a Randomized, Double-Blind, Placebo-Controlled Design After Single and Multiple Oral Dosing in Healthy Adult Volunteers
Brief Title: PK, Safety and Tolerability of Single and Multiple Doses of Oxfendazole Tablets
Acronym: HELP-OFZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Institute (Other); Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P1773-20A
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Filariasis
Keywords: Onchocerciasis; Parasitic Diseases; Neglected Disease; Phase I; Safety; Tolerability; Pharmacokinetics; Bioavailability; Volunteers
MeSH Terms: conditions — Filariasis; Onchocerciasis; Parasitic Diseases; Neglected Diseases | interventions — oxfendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Dose of 100mg Oxfendazole versus Placebo (Experimental): 8 participants will receive a single oral dose of 100mg of oxfendazole. 2 participants will receive a single oral dose of placebo.
  Interventions: Drug: Oxfendazole; Drug: Placebo
- Single Dose of 400mg Oxfendazole versus Placebo (Experimental): 8 participants will receive a single oral dose of 400mg of oxfendazole. 2 participants will receive a single oral dose of placebo.
  Interventions: Drug: Oxfendazole; Drug: Placebo
- Multiple Doses of 400mg Oxfendazole versus Placebo (Experimental): 8 participants will receive multiple oral doses of 400mg of oxfendazole on 5 consecutive days.
  2 participants will receive multiple oral doses of placebo on 5 consecutive days.
  Interventions: Drug: Oxfendazole; Drug: Placebo

INTERVENTIONS:
Drug: Oxfendazole — Oxfendazole is a benzimidazole anthelminthic drug.
Drug: Placebo — The placebo tablet is made using the same non-active ingredients and matches the investigational tablet.

SUMMARY:
The study evaluates the pharmacokinetics (PK), safety and tolerability of oxfendazole, after administration as a tablet formulation in healthy male and female participants.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double blinded, single center phase I bioavailability study with two Single Dose cohorts and one Multiple Doses cohort in a total of 30 healthy male and female healthy volunteers (10 per cohort).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and non-pregnant (confirmed by pregnancy test) and non-breastfeeding female participants (18 to 45 years of age at the time of consent).
* Willingness to give written consent to participate in the trial, after reading the participant information and consent form and after having had the opportunity to discuss the trial with the Investigator or any delegate.
* Ability to read and write and to understand the participant information sheet and the nature of the trial and any hazards from participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial.
* Women of childbearing potential (WOCBP) must agree to use a highly effective form of contraception in combination with a barrier method from at least 28 days prior to first dosage to 30 days after last dosage.
* Male participants must be willing to ensure the use of condoms from the first dosage to 90 days after last dosage.
* Normal body weight range (body mass index (BMI) between 18 and 29.9 kg/ m2)

Exclusion Criteria:

* Participation in another clinical trial within 3 months prior to the study, or within 5-times the half-life of the drug tested in the previous clinical trial, whichever is longer. (Time calculated relative to the last dose in the previous clinical trial).
* Regular daily consumption of more than one liter of xanthine-containing beverages (e.g. chocolates, tea, coffee or cola drinks).
* Regular daily consumption of more than 5 cigarettes daily.
* Use of a prescription medicine during the 28 days before the first dose of trial medication or use of an over-the-counter medicine, during the 7 days before the first dose of trial medication.
* Use of dietary supplements or herbal remedies (such as St John's Wort) known to interfere with the CYP3A4 and/or P-gp metabolic pathway during the 28 days before the first dose of trial medication.
* Therapies which may impact on the interpretation of study results in the opinion of the Investigator.
* Medical, social condition, psychiatric disorder or occupational reasons that, in the judgment of the Investigator, is a contraindication to protocol participation, may impair the volunteer's ability to give informed consent or effectively participate in the study, may significantly increase the risk to the volunteer because of participation in the study or may impair interpretation of the study data.
* Blood pressure and heart rate in supine position at the screening examination outside one (or more) of the ranges 105-136 mm Hg systolic, 58-84 mm Hg diastolic; heart rate 56- 96 beats/min.
* Febrile illness within 1 week before the start of study treatment.
* History of relevant diseases of vital organs, of the central nervous system or other organs.
* Participants with a history of allergies, non-allergic drug reactions, adverse reaction to any drug, or multiple drug allergies.
* Participants with a hypersensitivity to the investigational drug, related benzimidazole compounds or the control agent and/ or to inactive constituents.
* Presence or history of drug or alcohol abuse in the last 10 years.
* Surgery (e.g. stomach bypass) or medical condition that might affect absorption of study drug taken orally.
* Clinically relevant abnormal medical history, concurrent medical condition, acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous.
* Relevant pathological abnormalities in the ECG such as a second or third-degree atrioventricular (AV) block, prolongation of the QRS complex over 120 msec or of the QTcF-interval over 450 msec (corrected interval according to Fridericia's formula).
* Positive test for hepatitis B or C.
* Positive test for HIV.
* Positive pregnancy test (WOCBP).
* Positive stool or urine test for helminth infestation by Kato-Katz, urine filtration or Baermann test.
* Positive for malaria by thick blood smear.
* Positive test for (neuro-) cysticercosis.
* Positive test for echinococcosis.
* Positive test for onchocerciasis.
* Presence of abnormal physical findings, ECG, or laboratory values at the screening assessment that could interfere with the objectives of the trial or the safety of the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration curve from time zero to the last quantifiable concentration at time t (AUC0-t) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 48 hours after single dose administration
  For single dose arms
Area under the plasma concentration curve (AUC) from time zero extrapolated to infinity (AUC0-∞) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 48 hours after single dose administration
  For single dose arms
Maximum observed concentration (Cmax) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 48 hours after single dose administration
  For single dose arms
Time to maximum observed concentration (Tmax) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 48 hours after single dose administration
  For single dose arms
Elimination half-life (t1/2) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 48 hours after single dose administration
  For single dose arms
Area under the plasma concentration curve over dosing interval (AUCtau) of oxfendazole and its metabolites fenbendazole | At different time points from pre-dose up to 72 hours after last dose administration
  For multiple doses arm
Accumulation Ratio (Racc) of oxfendazole and its metabolites fenbendazole | At different time points from pre-dose up to 72 hours after last dose administration
  For multiple doses arm
Maximum observed concentration (Cmax) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 72 hours after last dose administration
  For multiple doses arm
Time to maximum observed concentration (Tmax) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 72 hours after last dose administration
  For multiple doses arm
Elimination half-life (t1/2) of oxfendazole and its metabolites fenbendazole and fenbendazole sulfone | At different time points from pre-dose up to 72 hours after last dose administration
  For multiple doses arm

SECONDARY OUTCOMES:
Safety and tolerability of oxfendazole as measured by number of participants with treatment related adverse events and serious adverse events | From Day 1 to Day 14.
  Number of participants with treatment related adverse events and serious adverse events
Safety and tolerability of oxfendazole as measured by number of participants with physical examination findings | At different time points from baseline to Day 14
  Number of participants with physical examination findings. Standard examination done on skin, lymph nodes, head, eyes, ears, nose, throat, respiratory, cardiovascular, abdomen, extremities, musculoskeletal, and neurological.
Safety and tolerability of oxfendazole as measured by number of participants with vital signs findings | At different time points from baseline to Day 14
  Number of participants with vital signs findings (heart rate, blood pressure, axillar temperature, respiratory rate,)
Safety and tolerability of oxfendazole as measured by number of participants with clinical laboratory test findings | At different time points from baseline to Day 14
  Number of participants with relevant abnormal clinical laboratory tests results (hematology (hemoglobin, white blood cells (differentiation of eosinophils and neutrophils) and platelets), coagulation (prothrombin time and activated partial thromboplastin time), biochemistry (Creatinine, Alanine aminotransferase, Aspartate aminotransferase, total bilirubin, sodium, potassium, chloride, bicarbonate, blood urea nitrogen), urinalysis (proteinuria and glucose))
Safety and tolerability of oxfendazole as measured by number of participants with 12-lead ECG findings Safety and tolerability of oxfendazole as measured by the change in ECG parameters | Pre-dose, 1 and 2 hours after single dose administration on Day 1; Pre-dose, 1 and 2 hours after dose administration on Day 1 and pre-dose, 1 and 2 hours after dose administration on Day 5 (last dose) for multiple doses administration arm.
  Number of participants with 12-lead ECG findings (heart rate (HR), PR interval, QRS, QT, QTcB, QTcF, cardiac rhythm and T wave morphology)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Paris, Study Director — Swiss TPH; Said Jongo, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided
It is intended that Summary results will be shared once Clinical Study Report will be available.

REFERENCES:
- [Derived] Assmus F, Adehin A, Hoglund RM, Nyaulingo G, Mbarak H, Jongo S, Ackermann E, Reus E, Keiser J, Rocha FBDS, Specht S, Scandale I, Tarning J. Repurposing Oxfendazole for Onchocerciasis: Population Pharmacokinetics of a Tablet Formulation in Healthy African Adults. CPT Pharmacometrics Syst Pharmacol. 2026 Feb;15(2):e70189. doi: 10.1002/psp4.70189. PMID 41662151